CLINICAL TRIAL: NCT06729021
Title: Predictive Efficacy of Modified Caprini Score and D-Dimer for the Evaluation and Management of Lower Extremity Venous Thrombosis Among Cardiothoracic Surgery Patients in Baghdad
Brief Title: Predictive Value of Modified Caprini Score and D-Dimer in Managing Lower Limb Venous Thrombosis in Cardiothoracic Patients
Acronym: DVT
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241207
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: DVT - Deep Vein Thrombosis
Keywords: Caprini Score; D-Dimer; DVT
MeSH Terms: conditions — Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: GCS — Graduated compression stockings may be used after procedure by the decision of the doctor
Drug: LMWH — Low-molecular-weight heparin may be used after procedure by the decision of the doctor

SUMMARY:
The goal of this observational study is to evaluate the predictive efficacy of the Modified Caprini Risk Assessment Score and D-Dimer in identifying and managing lower extremity venous thrombosis (LEVT) among cardiothoracic surgery patients in Baghdad. The main questions it aims to answer are:

Does combining the Modified Caprini Score with D-Dimer improve the accuracy of predicting lower extremity venous thrombosis (LEVT) compared to using each tool independently? Can these tools effectively guide clinical decisions for lower extremity venous thrombosis (LEVT) prevention and management in this patient population?

Participants will:

Undergo risk assessment for lower extremity venous thrombosis (LEVT) using the Modified Caprini Score and have their D-Dimer levels measured during their hospital stay.

Be monitored for clinical outcomes, including confirmed lower extremity venous thrombosis (LEVT) incidence, need for anticoagulation therapy, and complications such as pulmonary embolism or recurrent thrombosis.

DETAILED DESCRIPTION:
Research indicates that the incidence of deep vein thrombosis (DVT) among surgical patients is notably higher than in the general population. In a review of 10,638 cardiac surgical patients, the incidence of deep vein thrombosis (DVT) was found to be 0.7% due to multiple factors, including prolonged immobility, the hypercoagulable state induced by surgical interventions, and vascular trauma associated with cardiothoracic procedures. Patients undergoing cardiac surgery may have longer hospital stays, which correlates with increased risk for deep vein thrombosis (DVT). For instance, studies indicate that the incidence of deep vein thrombosis (DVT) in patients post-cardiac surgery can be as high as 1.62%. Certain surgeries, such as coronary artery bypass grafting (CABG) and valve surgeries, have shown a higher incidence of deep vein thrombosis (DVT) compared to other surgical procedures. For example, one study found that 1.62% of patients developed deep vein thrombosis (DVT) after cardiac surgery. Procedures like thoracotomy or pneumonectomy are associated with even higher risks due to the extensive surgical trauma involved. Research has indicated that patients undergoing such surgeries may experience DVT rates as high as 34.1%.

Lower extremity venous thrombosis (LEVT) is a significant clinical concern that encompasses deep vein thrombosis (DVT) and pulmonary embolism (PE) and poses a considerable risk postoperatively. The risk of PE is especially pronounced during the first six weeks post-surgery, with studies indicating that patients are up to 70 times more likely to experience VTE during this period compared to those who have not undergone surgery The risk remains elevated beyond six weeks, albeit at a reduced level. For instance, the odds ratio for PE between weeks 7 and 12 post-surgery can be as high as 4.23 for certain surgical types. This condition represents a continuum of pathology that can lead to severe outcomes, including sudden death from PE, This is considered one of the more serious postoperative complications. Early identification and the timely use of preventive measures can prevent PE and other fatal complications.

The extensive research currently conducted on the risk factors for postoperative VTE has yielded several risk assessment models. The Caprini score is widely used across various surgical specialties to identify patients at high risk of developing VTE. Among these, the modified Caprini score is the most commonly used tool in the thoracic surgery department. D-dimer is a biomarker of fibrin formation and degradation and acts a marker of coagulation and fibrinolysis system activation. As an indirect marker of thrombosis activity, D-dimer is of great significance for checking the formation of acute venous thrombosis. Although D-dimer has high negative predictive value for DVT, it has low positive predictive value and low specificity for thrombosis The Caprini score has been validated across numerous specialties in Iraq, confirming its reliability as a predictive tool for VTE. Many hospitals in Iraq lack modern medical equipment and resources that are essential for diagnosing and treating VTE effectively. This deficiency contributes to a reliance on outdated practices and guidelines, which may not align with current best practices in VTE management The slow adoption of new technologies impedes the ability to perform accurate risk assessments and implement evidence-based protocols for VTE prophylaxis. For instance, studies indicate that healthcare providers often depend on clinical experience rather than established guidelines due to a lack of access to updated resources The aim of this study is to bridge these gaps by investigating the efficacy of using a combined approach involving the modified Caprini risk assessment score and D-dimer testing values in patients with lower extremity venous thrombosis following cardiothoracic surgery We hypothesized that the combination of these two indicators may provide better predictive value. These findings may provide the basis for the follow-up prediction and timely intervention of high-risk groups of post-surgery patients, potentially leading to better patient outcomes. This combination approach has been explored in several international studies, but its application within Iraq, specifically in Baghdad, has yet to be thoroughly examined in cardiothoracic patients.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with a hospital stay over 3 days
* Written informed consent obtained from patients or their legal guardians.
* Availability for postoperative follow-up to assess outcomes like LEVT development or related complications.

Exclusion Criteria:

* Preexisting LEVT or Pulmonary Embolism: Diagnosed before the index surgery.
* Severe Coagulopathy: Patients with inherited or acquired bleeding disorders (e.g., hemophilia, advanced liver disease).
* receiving any anticoagulation therapy for any reason.
* patients who did not undergo a postoperative D-dimer test.
* Incomplete Data: missing essential clinical or laboratory data for Modified Caprini Score calculation or D-Dimer measurement.
* Pregnancy: pregnant women or those within six weeks postpartum.
* Noncompliance: Patients unwilling or unable to adhere to study follow-up protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients (≥18 years old) undergoing cardiothoracic surgery at Kadhimiya Teaching Hospital in Baghdad, with a focus on those at risk for lower extremity venous thrombosis (LEVT).
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
any episode of VTE (Venous Thromboembolism) | In-Hospital Phase (average of 7 days through discharge); Post-Discharge Follow-Up: Day 7, Day 15, and Day 30
  symptomatic or asymptomatic, confirmed by instrumental diagnostics.
Caprini risk assessment model scores | Day 1 preoperative (one day prior to surgery)
  rini risk assessment model scores were used to stratify patients into three groups: low risk (0-4 points), intermediate risk (5-8 points), and high risk (≥9 points)
Concentration of D-dimer in Blood Samples | Day 1 postoperative (the first day after surgery)
  The upper normal value 0.55mg/L FEU was used.

SECONDARY OUTCOMES:
Number of Participants with Symptomatic Pulmonary Embolism | In-Hospital Phase (average of 7 days through discharge); Post-Discharge Follow-Up: Day 7, Day 15, and Day 30
  symptomatic pulmonary embolism confirmed by perfusion isotope scanning or CT pulmonary angiography.
Recurrent Deep Vein Thrombosis (DVT) | Post-Discharge Follow-Up: Day 7, Day 15, and Day 30
  A new episode of deep vein thrombosis occurs after the initial diagnosis with clinical symptoms (such as leg pain, swelling, redness, or tenderness) and is confirmed through instrumental diagnostics (e.g., ultrasound, CT venography, MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Yaser aamer Eisa Alhaibi, Assistant professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mikhael, E.M., et al., Effectiveness of Pharmacist-Led Nurse Education on Enoxaparin Injection Technique in Baghdad Teaching Hospital, Iraq. Al-Rafidain J Med Sci, 2024. 6(1): p. 202207.
- [Background] Kareem, G.N. and S.K. Alalaf, Risk assessment and compliance with hospital guidelines for venous thromboprophylaxis after gynecological surgeries. Zanco J Med Sci, 2022. 26(2): p. 108-117.
- [Background] Weitz JI, Fredenburgh JC, Eikelboom JW. A Test in Context: D-Dimer. J Am Coll Cardiol. 2017 Nov 7;70(19):2411-2420. doi: 10.1016/j.jacc.2017.09.024. PMID 29096812
- [Background] Caprini JA. Thrombosis risk assessment as a guide to quality patient care. Dis Mon. 2005 Feb-Mar;51(2-3):70-8. doi: 10.1016/j.disamonth.2005.02.003. No abstract available. PMID 15900257
- [Background] Khan F, Tritschler T, Kahn SR, Rodger MA. Venous thromboembolism. Lancet. 2021 Jul 3;398(10294):64-77. doi: 10.1016/S0140-6736(20)32658-1. Epub 2021 May 10. PMID 33984268
- [Result] Almurshedi, I.M.K., A.M. Kamil, and A.A. Noaman, Evaluation of Risk Factors of Venous Thromboembolism in Imam Sadiq Teaching Hospital at Babylon City. Journal of Techniques, 2022. 4(Special Issue): p. 58-63.
- [Result] Suker SEJ, Al-Meen AAH, Khawwam AA. Assessment of knowledge and practice of venous thromboembolism (VTE) prophylaxis after cesarean section among gynecologists and obstetricians in Al-Najaf hospitals. J Med Life. 2021 Sep-Oct;14(5):690-694. doi: 10.25122/jml-2021-0226. PMID 35027972
- [Result] Alhilali, D.N., A. Tukmagi, and H.M. Abass, Venous thromboembolism risk and prophylaxis in hospitalized patients in Iraq. J Pharm Biomed Sci, 2016. 6: p. 2016
- [Result] Stender MT, Frokjaer JB, Hagedorn Nielsen TS, Larsen TB, Lundbye-Christensen S, Elbrond H, Thorlacius-Ussing O. Combined use of clinical pre-test probability and D-dimer test in the diagnosis of preoperative deep venous thrombosis in colorectal cancer patients. Thromb Haemost. 2008 Feb;99(2):396-400. doi: 10.1160/TH07-06-0397. PMID 18278191
- [Result] Abolfotouh MA, Almadani K, Al Rowaily MA. Diagnostic Accuracy of D-Dimer Testing and the Revised Geneva Score in the Prediction of Pulmonary Embolism. Int J Gen Med. 2020 Dec 15;13:1537-1543. doi: 10.2147/IJGM.S289289. eCollection 2020. PMID 33363402
- [Result] Ke L, Cui S, Yang M, Chen J, Xu S, Jiang G, Zhang Y, Chen S, Zheng E, Zhao H, Fan X, Li Y, Zhi X, Hu B, Li H; China Embolism-Thrombosis After Surgery of Thorax (ChEST) Study Group. Validation of a modified Caprini risk assessment model in lung cancer patients undergoing surgery: Results of a multicenter cross-sectional observational study. J Surg Oncol. 2022 Apr;125(5):933-942. doi: 10.1002/jso.26794. Epub 2022 Jan 18. PMID 35041203
- [Result] Caron A, Depas N, Chazard E, Yelnik C, Jeanpierre E, Paris C, Beuscart JB, Ficheur G. Risk of Pulmonary Embolism More Than 6 Weeks After Surgery Among Cancer-Free Middle-aged Patients. JAMA Surg. 2019 Dec 1;154(12):1126-1132. doi: 10.1001/jamasurg.2019.3742. PMID 31596449
- [Result] Sweetland S, Green J, Liu B, Berrington de Gonzalez A, Canonico M, Reeves G, Beral V; Million Women Study collaborators. Duration and magnitude of the postoperative risk of venous thromboembolism in middle aged women: prospective cohort study. BMJ. 2009 Dec 3;339:b4583. doi: 10.1136/bmj.b4583. PMID 19959589
- [Result] Fei W, Jian Z, Zhi G, Rong W, Jianxin L, Yongquan G, Weiping W. Analysis of risk factors for venous thromboembolism in patients after thoracic surgery: A clinical study of 167 cases. Turk Gogus Kalp Damar Cerrahisi Derg. 2018 Jan 9;26(1):93-98. doi: 10.5606/tgkdc.dergisi.2018.14980. eCollection 2018 Jan. PMID 32082717
- [Result] Khoury H, Lyons R, Sanaiha Y, Rudasill S, Shemin RJ, Benharash P. Deep Venous Thrombosis and Pulmonary Embolism in Cardiac Surgical Patients. Ann Thorac Surg. 2020 Jun;109(6):1804-1810. doi: 10.1016/j.athoracsur.2019.09.055. Epub 2019 Nov 7. PMID 31706868
- [Result] DeLaria GA, Hunter JA. Deep venous thrombosis. Implications after open heart surgery. Chest. 1991 Feb;99(2):284-8. doi: 10.1378/chest.99.2.284. PMID 1989784